CLINICAL TRIAL: NCT05329714
Title: PVRI Global Deep Phenotyping Meta-Registry for Pulmonary Hypertension
Brief Title: PVRI GoDeep Global Deep Phenotyping Meta-Registry for Pulmonary Hypertension
Acronym: PVRI GoDeep
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Imperial College London (Other); Johns Hopkins University (Other); Stanford University (Other); University of Sheffield (Other); University of Pittsburgh (Other); University of Pavia (Other); Hospital de Niños de la Santísima Trinidad (Unknown); Academy of Medical Sciences of Ukraine (Other); The Methodist Hospital Research Institute (Other); Vanderbilt University Medical Center (Other); Mayo Clinic (Other); National and Kapodistrian University of Athens (Other); Aristotle University Of Thessaloniki (Other); University Hospital of Targu Mures, Romania (Other); University Hospital Heidelberg (Other); Milpark Hospital (Unknown); University of Minnesota (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Fiona Stanley Hospital (Other); Sunshine Coast University Hospital (Unknown); China-Japan Friendship Hospital (Other); Medical University of Graz (Other); National Hospital Organization Okayama Medical Center (Other); Royal Hobart Hospital (Other Government); University Hospital, Zürich (Other); Universidad Nacional de La Plata (Other); Gold Coast Hospital and Health Service (Other Government)
Responsible Party: Sponsor
Other Study IDs: PVRIGoDeep
Record Dates: First submitted 2022-03-14; First posted 2022-04-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension; Global Health
Keywords: Pulmonary Hypertension; Data Integration; Standardization; Global Health; Quality Indicators
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Pulmonary Hypertension: Patients with a diagnosis of pulmonary hypertension typically diagnosed via right heart catheterization.
- Control Group: Participating PH centers can optionally provide data about patients with exclusion of pulmonary hypertension

SUMMARY:
PVRI-GoDeep is a PH Meta-Registry, run under the umbrella of the Pulmonary Vascular Research Institute (PVRI). It merges anonymized PH patient related data from various local registries around the world run under the responsibility of PVRI members. It will be operated under the auspices of the University of Giessen/Giessen PH center. Combining deep phenotyping with worldwide outreach, PVRI-GoDeep aims to offer insights into specific geographical and ethnical profiles of PH, to deepen the epidemiological, clinical and molecular understanding of this disease and to promote strategies for improved individualized treatment of PH patients.

DETAILED DESCRIPTION:
PVRI-GoDeep is a PH Meta-Registry, run under the umbrella of the Pulmonary Vascular Research Institute (PVRI). It merges anonymized PH patient related data from various local registries around the world run under the responsibility of PVRI members. It will be operated under the auspices of the University of Giessen/Giessen PH center.

Combining deep phenotyping with worldwide outreach, PVRI-GoDeep aims to offer insights into specific geographical and ethnical profiles of PH, to deepen the epidemiological, clinical and molecular understanding of this disease and to promote strategies for improved individualized treatment of PH patients.

The data provided by PVRI-GoDeep will support academia to perform scientific projects in the field of PH. Pharmaceutical / commercial companies will be charged fee for access to PVRI-GoDeep data and / or analysis, thereby creating revenues exclusively devoted to support the PVRI mission and the registries entering their data into PVRI-GoDeep. All requests from academia or commercial companies are to be decided by the PVRI-GoDeep consortium, serving as Use and Access Committee.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Pulmonary Hypertension

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Global cohort of patients with pulmonary hypertension (PH)
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2050-01-30 (Estimated); Study Completion 2055-01-30 (Estimated)

PRIMARY OUTCOMES:
Global analysis of PH patients | From entry into the registry up to 10 years
  Global comparison and analysis of the course of disease of PH patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Giessen PH Center, Giessen, Hesse, Germany

REFERENCES:
- [Derived] Yogeswaran A, Gall H, Funderich M, Wilkins MR, Howard L, Kiely DG, Lawrie A, Hassoun PM, Sirenklo Y, Torbas O, Sweatt AJ, Zamanian RT, Williams PG, Frauendorf M, Arvanitaki A, Giannakoulas G, Saleh K, Sabbour H, Cajigas HR, Frantz R, Al Ghouleh I, Chan SY, Brittain E, Annis JS, Pepe A, Ghio S, Orfanos S, Anthi A, Majeed RW, Wilhelm J, Ghofrani HA, Richter MJ, Grimminger F, Sahay S, Tello K, Seeger W; Pulmonary Vascular Research Institute GoDeep Consortium. Comparison of Contemporary Risk Scores in All Groups of Pulmonary Hypertension: A Pulmonary Vascular Research Institute GoDeep Meta-Registry Analysis. Chest. 2024 Sep;166(3):585-603. doi: 10.1016/j.chest.2024.03.018. Epub 2024 Mar 19. PMID 38508334